CLINICAL TRIAL: NCT05616845
Title: A mHealth Application as a Screening Tool for Neonatal Jaundice in Filipino Neonates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Picterus AS (Industry)
Collaborators: Norwegian University of Science and Technology Faculty of Medicine and Health Sciences Department of Public Health and Nursing (Unknown); Gov. Celestino Gallares Memorial Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 322016
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2022-11-23 (Actual); Status verified 2022-11

CONDITIONS: Jaundice, Neonatal
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Enable high qualitative estimation of bilirubin levels in the blood of new-borns (Experimental): There is only one arm in this study which is to enable high qualitative estimation of bilirubin levels in the blood of new-borns with darker skin and with high melanin content such as Filipino neonates.
  Interventions: Device: Picterus Jaundice Pro

INTERVENTIONS:
Device: Picterus Jaundice Pro — Use Picterus Jaundice Pro, a smartphone app that is used to take photo of the newborns skin, where the Picterus calibration card is place.
  Other Names: Picterus JP

SUMMARY:
The purpose of the study is to test the reliability of the Picterus smartphone application in Filipino neonates. A descriptive cross-sectional study will be the method to understand the correlation of the modalities and to determine the reliability of the application

DETAILED DESCRIPTION:
The purpose of the study is to test the reliability of the Picterus smartphone application.

The study is designed for Filipino neonates, but implemented in other LMIC. The participants include newborns with or without jaundice, Gestational age >37 weeks, Age0-14days, Weight >2500 gram and absence of congenital malformations. Demographic data of the neonates will be collected together with all the performed tests and it will be stored in a secured system. Blood will be drawn and measure the bilirubin level of the neonates in a standard clinical routine and will be compared to the estimated bilirubin performed with the Picterus smartphone application.

A descriptive cross-sectional study will be the method to understand the correlation of the modalities and to determine the reliability of the application.

It will provide an answer to whether the Picterus smartphone application is reliable to other populations, especially to darker skin and with high melanin content such as Filipino neonates.

ELIGIBILITY:
Inclusion Criteria:

* Newborns with or without jaundice
* Gestational age ≥ 37 weeks
* Age 0 - 14 days
* Weight 2500 to 4500 grams
* Absence of congenital malformations

Exclusion Criteria:

* Newborns with life-threatening conditions or significant illness

  * Newborns diagnosed with inborn errors of metabolism
  * Jaundiced newborns that have undergone phototherapy before screening

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 69 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-02-26 (Actual)

PRIMARY OUTCOMES:
validate the reliability of the Picterus mHealth application as a screening tool for neonatal jaundice in Filipino neonates | 5-10 minutes
  Validation of smartphone-based screening tool (Picterus JP) for neonatal jaundice in newborns with high melanin content.

SECONDARY OUTCOMES:
correlation between the estimated levels of bilirubin detected by the Picterus mHealth application and bilirubin serum levels in Filipino neonates | 1-2 hours
  correlation between the estimated levels of bilirubin detected by the Picterus mHealth application and bilirubin serum levels in Filipino neonates
correlation between the estimated level of bilirubin detected by the Picterus mHealth application and transcutaneous bilirubinometer results in Filipino neonates. | 5-10 minutes
  correlation between the estimated level of bilirubin detected by the Picterus mHealth application and transcutaneous bilirubinometer results in Filipino neonates.
correlation between the estimated level of bilirubin detected by the Picterus mHealth application and those obtained using visual Kramer scale in Filipino neonates. | 5 minutes
  correlation between the estimated level of bilirubin detected by the Picterus mHealth application and those obtained using visual Kramer scale in Filipino neonates.
sensitivity, specificity, positive and negative predictive value between estimated bilirubin level of the digital images, Kramer examination and TcB. | 5 months
  sensitivity, specificity, positive and negative predictive value between estimated bilirubin level of the digital images, Kramer examination and TcB.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Øyvind Odland, Prof,MD,PhD, Study Director — NTNU Faculty of Medicine and Health Sciences, Department of Public Health and Nursing
Locations (1):
- Governor Celestino Gallares Memorial Hospital, Tagbilaran City, Bohol, Philippines

REFERENCES:
- See also: Master thesis describing the study and its results — https://ntnuopen.ntnu.no/ntnu-xmlui/handle/11250/3006144